CLINICAL TRIAL: NCT02833194
Title: Assessment of the Prevalence of Major Psychiatric Disorders in a Cohort of Women With Clinical Criteria Corresponding to Pure, Abortive-form, Obstetrical, Antiphospholipid Syndrome
Acronym: NOHA-PSY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/JCG-01
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2023-06

CONDITIONS: Antiphospholipid Syndrome; Factor V Leiden Thrombophilia
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombophilia due to Activated Protein C Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Leiden Group: Women with an isolated F5 rs6025 polymorphism or an isolated F2 rs1799963 polymorphism.
- aP1Ab-positive: Inclusion in the "aP1Ab" Group:
  * Initially positive for aP1Ab
  * Second positive aP1Ab test six months later
- Thrombophilia-negative: Women with completely negative thombophilia screening results.

SUMMARY:
The primary objective of this study was to evaluate and compare the prevalence of the following psychiatric pathologies (based on the MINI5.0.0 questionnaire) among 3 groups of women (Leiden versus aP1Ab-positive versus thrombophilia-negative) with similar obstetrical histories 10 years after their initial assessment/diagnosis.

* Mood disorders, including depressive episodes during the previous two weeks, recurrent depressive disorders at any point in life, dysthymia in the last two years, or any current or past manic episode;
* Anxiety disorders, including current agoraphobia, current panic disorders, agoraphobia with panic disorders, current social phobia, generalized anxiety in the last 6 months, or current posttraumatic stress syndrome;
* Apparent psychotic syndromes, including isolated or recurrent psychotic syndromes, past or present (clinically validated),
* Current alcohol or drug problems (dependence or abuse).

ELIGIBILITY:
Inclusion Criteria:

* Three unexplained consecutive spontaneous abortions before the 10th week of gestation (the recurrent embryo loss subgroup) - OR -
* One unexplained death of a morphologically normal fetus (fetal loss) at or after the 10th week of gestation (fetal loss subgroup).

Exclusion Criteria:

* Any history of thrombotic events or any treatment given during previous pregnancies that might have modified the natural course of the condition
* Women whose pregnancy losses could be explained by infectious, metabolic, anatomic or hormonal facotrs, or associated with paternal or maternal chromosomal causes
* Seropositivity for HIV, hepatitis B or C
* Women with antithrombin, protein C, or protein S deficiency, and women with abnormal fibrinogen or with the JAK2 V617F mutation were further excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were selected via the regional NOHA (Nîmes Obstetricians and Hematologists - Antiphospholipid Syndrome study) network, which referred women with losses of spontaneous pregnancies to the Hematology Outpatient Department of the Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1592 (Actual)
Dates: Start 2005-07; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mini Internationl Neuropsychiatric Interview 5.0.0 | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Gris JC, Cyprien F, Bouvier S, Cochery-Nouvellon E, Lavigne-Lissalde G, Mercier E, Balducchi JP. Antiphospholipid antibodies are associated with positive screening for common mental disorders in women with previous pregnancy loss. The NOHA-PSY observational study. World J Biol Psychiatry. 2019 Jan;20(1):51-63. doi: 10.1080/15622975.2017.1333146. Epub 2017 Jun 19. PMID 28532221